CLINICAL TRIAL: NCT00840944
Title: Efficacy and Safety of a 4 Year Combination Therapy of Growth Hormone and Gonadotropin- Releasing Hormone Agonist in Children With a Short Predicted Height.
Brief Title: A 4 Year Combination Therapy of Growth Hormone and (GnRH) Agonist in Children With a Short Predicted Height
Acronym: ZomaTrip
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belgian Study Group for Pediatric Endocrinology (Other)
Responsible Party: Principal Investigator, Hilde Dotremont, MD, Belgian Study Group for Pediatric Endocrinology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2007-003247-70
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Idiopathic Short Stature
Keywords: gonadotropin releasing hormone agonist; growth hormone; final height; bone density; puberty
MeSH Terms: interventions — Human Growth Hormone; Growth Hormone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZOMATRIP (Experimental): GnRH agonist triptorelin plus somatropin
  Interventions: Drug: somatropin; Drug: triptorelin

INTERVENTIONS:
Drug: somatropin — somatropin 0.050 mg/kg/day
  Other Names: growth hormone; zomacton
Drug: triptorelin — triptorelin 3.75 mg each month
  Other Names: decapeptyl

SUMMARY:
Estrogens are responsible for the disappearance of growth cartilage in the long bones at the end of the pubertal growth spurt both in boys and in girls. It is therefore hypothesized that stopping pubertal development and hence estrogen production, will prolong and increase the pubertal growth spurt, especially when growth hormone is given concommitantly.

Boys in early puberty, with a bone age between 11 and 13 years and a predicted adult height below 163 cm or girls in early puberty with a bone age between 10 and 12 years and a predicted height under 151 cm will be treated with triptorelin 3.75 mg and Zomacton growth hormone for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult height prediction below -2.5 SD : 151 cm for girls and 164 cm for boys based on the vlaamse groeicurve 2004 (vub.ac.be/groeicurven)
* Pubertal: breast development at least M2 for girls and at least 4 ml of testicular volume for boys
* Bone age >10 years but < 12 years for girls and > 11 but < 13 years for boys
* Signed informed consent

Exclusion Criteria:

* Adopted children ( different genetic background, lack of data on birth parameters and parents)
* Bone dysplasia or sitting height/ total height > 2 SDS on standards by Gerver et al (see appendix)
* Chronic use of glucocorticoids
* Previous growth promoting therapy such as GH, sex steroids, oxandrolone,
* Known GH deficiency
* Chronic infectious disease
* Active rheumatic disease
* Previously diagnosed or currently suspected malignancy
* Sex steroid therapy
* Diabetes mellitus
* Renal insufficiency (serum creatinine > 1.5 mg/dl)
* Hepatic disease ( liver test > 4 fold upper limit of normality)
* Current congestive heart failure
* Inability to follow the study protocol
* Treatment with a non registered drug during the last 30 days before the moment of inclusion.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
height | 6 - 8 years
  Difference between predicted height at start of treatment and adult height

SECONDARY OUTCOMES:
bone density | 6 - 8 years
  Bone density SDS measured by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Dotremont, MD, Principal Investigator — BSGPE
Locations (6):
- Belgium (6):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Jessah Ziekenhuis, Hasselt, Limburg
  - Kinderziekenhuis UGent, Ghent, Oost Vlaanderen
  - Hopital Universitaire Reine Fabiola (HUDERF), Brussels
  - Kinderziekenhuis UZ Brussel, Brussels
  - CHU ND-des Bruyères, Liège

REFERENCES:
- [Derived] Dotremont H, France A, Heinrichs C, Tenoutasse S, Brachet C, Cools M, De Waele K, Massa G, Lebrethon MC, Gies I, Van Besien J, Derycke C, Ziraldo M, De Schepper J, Beauloye V, Verhulst S, Rooman R, den Brinker M. Efficacy and safety of a 4-year combination therapy of growth hormone and gonadotropin-releasing hormone analogue in pubertal girls with short predicted adult height. Front Endocrinol (Lausanne). 2023 Mar 17;14:1113750. doi: 10.3389/fendo.2023.1113750. eCollection 2023. PMID 37008942